CLINICAL TRIAL: NCT05836363
Title: Fate at Long-term of Mild to Moderate Bicuspid Aortic Valve Disease Left Untreated at the Time of Supracoronary Ascending Aorta Replacement
Status: Completed | Type: Observational
Sponsor: Michele De Bonis (Other)
Responsible Party: Sponsor-Investigator, Michele De Bonis, Chief of Cardiac Surgery of the Advanced and Research Therapies, Ospedale San Raffaele
Organization: Ospedale San Raffaele (Other)
Other Study IDs: NO SVAO-BAV
Record Dates: First submitted 2023-01-30; First posted 2023-05-01 (Actual); Last update posted 2023-05-01 (Actual); Status verified 2023-04

CONDITIONS: Bicuspid Aortic Valve; Ascending Aorta Aneurysm
MeSH Terms: conditions — Bicuspid Aortic Valve Disease; Aneurysm, Ascending Aorta

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Ascending aorta replacement — The aneurysmatic ascending aorta tract is replaced with a tubular dacron prosthesis

SUMMARY:
Aortic valve bicuspid disease is the most common congenital heart disease. It affects 0.5-2% of the population and is associated with an increased risk of developing aortic or ascending aortic valve complications.

There is no agreement regarding the opportunity for a "prophylactic" simultaneous aortic valve replacement in the case of mild or moderate aortic valve disease in the bicuspid valve, in patients with an indication for replacement of the ascending aorta due to an aneurysm involving its supra-coronary tract.

The aim of this study is to evaluate the long-term evolution of mild and moderate aortic valve disease in untreated bicuspid valve during supracoronary ascending aortic replacement surgery at our institution.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients;
* Bicuspid aortic valve;
* Presence of ascending aortic aneurysm in the supra-coronary tract treated with replacement using a prosthetic tube between 2002 and January 2020;
* Untreated aortic valve disease of no more than moderate degree (<2+) at the time of ascending aorta surgery.

Exclusion Criteria:

* Emergency/urgency procedures;
* Presence of aneurysm extending to the aortic arch or aortic root, with indication for aortic root or aortic arch surgery;
* Tricuspid aortic valve tricuspid;
* Absence of aortic valve disease;
* Presence of moderate-severe or severe aortic valve disease, with indication to a concomitant aortic valve replacement.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with bicuspid aortic valve and supra-coronaric ascending aorta aneurysm requiring ascending aorta replacement. Aortic valve regurgitation is no more than moderate, so it is left untreated following the guidelines.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2020-12-04 (Actual); Primary Completion 2020-12-09 (Actual); Study Completion 2020-12-09 (Actual)

PRIMARY OUTCOMES:
Aortic valve regurgitation | Through study completion, a minimum of 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Ospedale San Raffaele, Milan, Italy

IPD SHARING:
Plan to Share IPD: No